CLINICAL TRIAL: NCT07159763
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of CD388, a Novel Long-Acting Antiviral Conjugate, for the Prevention of Influenza in Adults and Adolescents at Higher Risk of Developing Influenza Complications
Brief Title: A Study to Evaluate the Safety and Efficacy of CD388 for Prevention of Influenza
Acronym: ANCHOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CD388.SQ.3.06
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Influenza
Keywords: Influenza; Antiviral Agents
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CD388 (Experimental): Participants are randomized to receive 450 milligrams (mg) CD388 by SQ injection. Participants are randomized at a 1:1 ratio between the 2 arms.
  Interventions: Combination Product: CD388 Injection
- Placebo (Placebo Comparator): Participants are randomized to receive placebo by SQ injection. Participants are randomized at a 1:1 ratio between the 2 arms.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: CD388 Injection — CD388 liquid for injection
  Arms: CD388
Combination Product: Placebo — Placebo to match
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how well CD388 works in preventing symptomatic laboratory-confirmed influenza infections, as compared to placebo, when given as a single dose via 3 subcutaneous (SQ) injections to adult and adolescent participants who are at higher risk of developing influenza complications, and to evaluate the safety and tolerability of CD388, as compared to placebo.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy, safety, and tolerability of CD388 administered as a single dose via 3 SQ injections in adult and adolescent participants who are at higher risk of developing complications from influenza.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 12 years of age or older at the time of signing the informed consent.
2. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA] in the US) obtained from the participant before performing any protocol-related procedures, including screening evaluations. For participants under the legal age of consent as defined by local regulations, the parent(s) or legal guardian(s) may be required to give their signed written informed consent and participants may sign an assent form as specified by local law.
3. Has negative rapid antigen tests for influenza and severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) prior to dosing at Day 1.
4. Weight is ≥ 40 kilograms (kg) at screening.
5. Body Mass Index (BMI; calculated as weight in kg divided by height in meters [m] squared)) is ≥ 18 kg/m^2 at screening.
6. In the opinion of the Investigator, must be able to comply with the requirements of the protocol and be able to read, understand, and complete questionnaires in the electronic diary (eDiary), work with smartphones/tablets/computers (if applicable, with assistance by a caregiver, surrogate, or legally authorized representative), and be willing and able to adhere to the prohibitions and restrictions specified in this protocol. If an appropriate language version is not available for the eDiary assessments, the participant should not be enrolled.
7. Must be assessed by the Investigator as medically stable and not requiring significant change in maintenance therapy and has not been hospitalized for worsening disease or any significant medical event during the 2 months before screening
8. Must agree to the following contraception requirements:

   a. Females of childbearing potential must use a highly effective, preferably user-independent, method of contraception (failure rate of less than 1 percent per year when used consistently and correctly) from ≥2 weeks prior to randomization and agree to remain on a highly effective method from Day 1 until 32 weeks after study intervention administration, the end of relevant systemic exposure. Note: A woman is considered of childbearing potential (i.e., fertile) following menarche and until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

   Note: Contraceptive (birth control) use by participants should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies.
9. Must agree not to donate blood or blood products from Day 1 until 32 weeks after study intervention administration.
10. Must be willing to provide verifiable identification, has means to be contacted, and is able to contact the Investigator/study site and communicate reliably during participation in the study.
11. In addition to inclusion criteria 1 through 10 above, participants are eligible to be included in Primary Stratum A of the study (higher risk non-immunocompromised) only if one or more of the following criteria apply:

    1. Has a history of pulmonary disease; specifically:

       * Chronic obstructive pulmonary disease (COPD), including chronic bronchitis and emphysema, graded as follows using the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Categories A, B, and E (ABE) (i.e., GOLD ABE) assessment tool:

         * Gold Grade 2 (moderate) or Grade 3 (severe) with following exacerbation history, within 1 year of screening

           * At least 2 moderate exacerbations (i.e., not leading to hospitalization), or
           * At least 1 exacerbation leading to hospitalization OR
         * Gold Grade 4 regardless of exacerbation history
       * Bronchiectasis, cystic fibrosis, interstitial lung disease, pneumoconiosis, or past or active bronchopulmonary dysplasia.
    2. Has moderate to severe asthma, as defined by the Global Initiative for Asthma (GINA) Treatment Steps 3-5.
    3. Has existing cardiac disease; specifically:

       * Congenital heart disease
       * Congestive heart failure New York Heart Association (NYHA) Class II-IV
       * Coronary artery disease requiring regular medication and/or follow-up for ischemic heart disease (i.e., participants who, through interventional procedure[s] and/or active medical treatment, have attained an established state of chronic stability of a duration of no less than 6 months)
       * Hypertension with cardiac complications (NOTE: Hypertension alone without cardiac complications will be excluded). Acceptable cardiac complications of hypertension include, but are not limited to, heart failure, cardiac arrhythmias (e.g., atrial fibrillation), ischemic heart disease, coronary artery disease, enlarged left heart, metabolic syndrome, left ventricular hypertrophy, systolic or diastolic myocardial dysfunction, angina, and myocardial infarction.
    4. Has insulin-dependent diabetes.
    5. Has moderate renal impairment (Stage 3 Chronic Kidney Disease [CKD], equivalent to an estimated glomerular filtration rate [eGFR] 30 to 59 milliliter per minute [mL/min] per 1.73 m^2 as calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation for adults or the Chronic Kidney Disease in Children under 25 [CKiD U25] equation for adolescents) with or without micro-macroproteinuria and within 3 months prior to screening; examples include, but are not limited to, any history of glomerulosclerosis, diabetic nephropathy, lupus nephritis, glomerular nephritis, immunoglobulin A (IgA) nephropathy, and Goodpasture syndrome. NOTE: Participants with chronic renal disease who meet the criteria for immune compromised (immunosuppressive therapy) should be enrolled in Stratum B.
    6. Is ≥ 65 years of age at the time of randomization but does not meet any of criteria 11a through 11e, and is otherwise healthy as determined by the Investigator.
12. In addition to inclusion criteria 1 through 10 above, participants are eligible to be included in Primary Stratum B of the study (immunocompromised) only if one or more of the following criteria apply:

    1. Has a solid tumor diagnosis AND has received chemotherapy and/or immunotherapy within 1 year of screening.
    2. Has a diagnosis of a hematologic malignancy within 5 years of screening AND has received any chemotherapy or biologic therapy within 1 year of screening.

       NOTE: Participants with multiple myeloma may be enrolled regardless of duration of time from diagnosis to screening.
    3. Participants who have had a solid organ transplant (SOT) must satisfy all of the following:

       * Has received a kidney, liver, heart, or lung transplant more than 6 months prior to screening
       * Is currently receiving at least two immunosuppressive medications
    4. Participants who have had a hematopoietic stem cell transplant (HSCT) must satisfy at least one of the following:

       * Has a history of HSCT (i.e., autologous, allogeneic, bone marrow, peripheral blood stem cell, tandem [peripheral blood and marrow]) within 1 year of screening
       * Has a history of non-autologous HSCT with graft-versus-host disease (GvHD) requiring active treatment with immunosuppressants (e.g., systemic corticosteroids ≥1 mg/kg at screening), regardless of the duration of time since HSCT
    5. Is receiving immunosuppressive medicines (e.g., corticosteroids [i.e., at least 20 mg prednisone or equivalent per day], alkylating agents, antimetabolites, transplant-related immunosuppressive drugs, cancer chemotherapeutic agents classified as severely immunosuppressive [e.g., Bruton's tyrosine kinase inhibitors], tumor- necrosis blockers, or other immunosuppressive biologic agents [e.g., for rheumatic diseases]). NOTE: The regimen must be stable (same agents and doses, or clinically equivalent doses) for ≥2 months prior to Screening to ensure clinical stability (see Inclusion Criterion 7).
    6. Has received chimeric antigen receptor-modified T-cell therapy.
    7. Has received B-cell depleting therapies (e.g., rituximab, ocrelizumab, ofatumumab, alemtuzumab) within the 12 months prior to screening.
    8. Has a diagnosis of any primary or secondary immunodeficiency except IgA deficiency.
    9. Has advanced or untreated human immunodeficiency virus (HIV) infection manifested by a cluster of differentiation 4 (CD4) cell count less than 350/cubic millimeter (mm^3) within 6 months of screening.

Exclusion Criteria:

1. A female who is pregnant or lactating.
2. Known or suspected allergy or history of anaphylaxis or other serious adverse reactions to zanamivir (following administration of inhaled or intravenous formulations), monoclonal antibodies (including crystallizable fragment [Fc] domains), or any of the components of CD388 or placebo.
3. Has been diagnosed with influenza (i.e., with medical history [including verbal] of influenza) within 6 months prior to randomization.
4. Has received the current seasonal inactivated influenza vaccine or live attenuated influenza vaccine within the 14 days prior to dosing on Day 1. (NOTE: Participant may have received recombinant influenza vaccine up to the day of dosing on Day 1.)
5. Has an acute (time-limited) or febrile (temperature ≥38.0 degrees Celsius [ºC] [≥100.4 degrees Fahrenheit {ºF}]) illness within 7 days prior to planned dosing on Day 1.
6. Has had close contact (including household contact) with someone with laboratory-confirmed influenza or SARS-CoV-2 or with someone who has been treated with antiviral therapies for influenza or SARS-CoV-2 within the 7 days prior to randomization.
7. Has a clinically unstable condition including, but not limited to, a psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior, or any other condition for which, in the opinion of the Investigator, may lead to hospitalization or death within the study period and that suggests that study enrollment would not be in the participant's best interest and/or that could prevent, confound, or limit the protocol-specified assessments.
8. Has any history of alcohol or drug abuse that, in the opinion of the Investigator, would adversely impact the conduct of the study.
9. Had major surgery (e.g., major cardiac, pulmonary or abdominal operation) within 4 weeks prior to randomization, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to participate in the study.
10. Has severe CKD (equivalent to an eGFR less than 30 mL/min/1.73 m^2 as calculated by CKD-EPI equation for adults or the CKiD U25 equation for adolescents), or is receiving hemodialysis.
11. Has screening electrocardiogram (ECG) findings of prolonged QT interval corrected using Fridericia's formula (QTcF) (greater than 450 milliseconds [msec] in males or greater than 470 msec in females), prolonged PR interval (greater than 220 msec), second- or third-degree heart block, or other clinically significant dysrhythmias, unless participant has a known cardiac diagnosis responsible for the ECG findings and is in stable condition. NOTE: Participants with cardiac pacemakers may be enrolled if no exclusion criteria are met.
12. Current or planned participation in another clinical study in which study intervention is being administered during participation in the current study. NOTE: Concurrent enrollment is allowed during the follow-up phase of the other clinical study or in case the study intervention in the other clinical study is a marketed product already approved for another indication - exception being if the other study requires study interventions that could affect the safety assessments of the present study (e.g., clinical laboratory tests).
13. Receipt within the past 30 days or 5 half-lives (whichever is longer) or anticipated receipt of any drug or other biologic agent (e.g., monoclonal antibodies) administered for the prevention or treatment of influenza.
14. Receipt of any formulation of immunoglobulin within 14 days prior to planned study intervention administration.
15. Receipt of any experimental drug, vaccine, or biologic agent within the 90 days or 5 half-lives (whichever is longer) prior to study intervention administration.
16. Has a clinically significant bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder) or medical history of significant bleeding or bruising following intramuscular or SQ injections or venipuncture. NOTE: Participants receiving apixaban or warfarin may be enrolled if the Investigator determines risk of SQ treatment with study intervention on Day 1 is minimal.
17. Has donated ≥450 mL of blood product (1 unit) for any reason within 30 days of screening.
18. Has direct involvement in the proposed study or other studies under the direction of the Investigator, sub-investigators, or at the study site; or is a family member of an individual with such direct involvement; or is an employee of the Sponsor; or was previously enrolled and dosed in a CD388 clinical trial.
19. In the Investigator's judgment, the participant has any condition or circumstance present that significantly increases risk, affects the ability to participate, impairs interpretation of study data, or indicates a likelihood of non-adherence to study requirements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Protocol-defined Influenza-like Illness (ILI) Occurring ≥7 Days after and up to 24 Weeks after Administration of Study Drug | From Day 8 up to 24 weeks after study drug dosing
  Percentage of participants experiencing protocol-defined ILI occurring after administration of CD388, with influenza infection confirmed by a reverse-transcriptase polymerase chain reaction positive (RT-PCR+) result based on a nasopharyngeal (NP) swab assayed at a central laboratory (first occurrence only), as compared to placebo.

SECONDARY OUTCOMES:
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) after Administration of Study Drug | From Day 1 through Day 197/End of Study (EOS) after study drug dosing
  Safety and tolerability of CD388, as compared to placebo, will be evaluated by assessing the number of participants with incidences of TEAEs following the administration of study drug. TEAEs include but are not limited to adverse events (AEs), serious adverse events (SAEs), injection site reactions (ISRs), and any potentially clinically significant changes from baseline seen in vital signs and clinical laboratory parameters.
Trough Plasma Concentration at 24 Weeks (C[trough24w]) Following Administration of CD388 | Based on sampling done at onsite visits on Day 8 (±3 days), Day 29 (±3 days), and Day 197/EOS (±7 days)
  Evaluation of the trough plasma concentration at 24 weeks (C[trough24w]) after study drug dosing.
Maximum Plasma Concentration (C[max]) Following Administration of CD388 | At onsite visits done on Day 8 (±3 days), Day 29 (±3 days), and Day 197/EOS (±7 days)
  Evaluation of the maximum plasma concentration (C[max]) after study drug dosing.
Area Under the Plasma Concentration-Time Curve (AUC) Following Administration of CD388 | At onsite visits done on Day 8 (±3 days), Day 29 (±3 days), and Day 197/EOS (±7 days)
  Evaluation of the area under the plasma concentration-time curve (AUC) after study drug dosing.
Detection of Anti-Drug Antibodies (ADAs) in Participants Administered CD388 | On Day 1 (pre-dose baseline) and at onsite visits done on Day 29 (±3 days) and Day 197/EOS (±7 days)
  Evaluation of blood serum samples for the detection of treatment-emergent anti-drug antibodies (ADAs) or treatment-boosted ADAs (based on an increase in ADA titer in samples positive for ADA at baseline) in participants administered CD388.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Davarpanah, MD, JD, Study Director — Cidara Therapeutics Inc.
Locations (150):
- United States (120):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - HOPE Research Institute, Glendale, Arizona
  - Desert Clinical Research, LLC / Avacare, Mesa, Arizona
  - Foothills Research Center / Avacare, Phoenix, Arizona
  - Fiel Family and Sports Medicine / Avacare, Tempe, Arizona
  - HOPE Research Institute, Tempe, Arizona
  - Arizona Clinical Trials, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Triallogix Medical Corporation, Fullerton, California
  - National Institute of Clinical Research, Inc., Garden Grove, California
  - Eximia Research-CA, LLC, La Mesa, California
  - Kinetic Clinical Research, LLC dba Long Beach Clinical Trials, Long Beach, California
  - Seaside Medical Group, Oceanside, California
  - Profound Research, LLC, Pasadena, California
  - Paradigm Clinical Research, Redding, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Acclaim Clinical Research, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Tekton Research, LLC, Denver, Colorado
  - Tekton Research, LLC, Fort Collins, Colorado
  - Critical Care, Pulmonary and Sleep Associates PLLP / Avacare, Lakewood, Colorado
  - Tekton Research, LLC, Longmont, Colorado
  - New England Research Associates, Bridgeport, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Imagine Research - Palm Beach County, Boynton Beach, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Hillcrest Medical Research, LLC, DeLand, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Flourish Research - Miami, LLC DBA Flourish Research, Miami, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Health Awareness, Inc., Port Saint Lucie, Florida
  - Global Clinical Professionals, St. Petersburg, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - DelRicht Research, Atlanta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Paradigm Clinical Research, Boise, Idaho
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Great Lakes Clinical Trials, LLC dba Flourish Research, Chicago, Illinois
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - Integrated Clinical Trial Services, LLC, West Des Moines, Iowa
  - Johnson County Clin-Trials, LLC, Lenexa, Kansas
  - AMR Clinical, Newton, Kansas
  - DelRicht Research, Louisville, Kentucky
  - Elevate Clinical Research, Lake Charles, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - Annapolis Internal Medicine / Avacare, Annapolis, Maryland
  - Jadestone Clinical Research, LLC, Silver Spring, Maryland
  - Skylight Health Research, Burlington, Massachusetts
  - Profound Research, LLC, Clarkston, Michigan
  - Profound Research, LLC, Dearborn, Michigan
  - Profound Research, LLC, Farmington Hills, Michigan
  - Javara, Inc., Mankato, Minnesota
  - DelRicht Research, Gulfport, Mississippi
  - Clay Platte Family Medicine, PC / Avacare, Kansas City, Missouri
  - DelRicht Research, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Methodist Physicians Clinic / Avacare, Fremont, Nebraska
  - Velocity Clinical Research - Omaha, Omaha, Nebraska
  - Midwest Regional Health Services, LLC / Avacare, Omaha, Nebraska
  - Henderson Clinical Trials, Henderson, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Santa Rosa Medical Centers of Nevada / Avacare, Las Vegas, Nevada
  - Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - IMA Clinical Research, Warren Township, New Jersey
  - Brooklyn Clinical Research, Brooklyn, New York
  - Finger Lakes Medical Research, PLLC dba Certified Research Associates, Cortland, New York
  - Drug Trials America, Hartsdale, New York
  - Rochester Clinical Research, Rochester, New York
  - CHEAR Center, LLC, The Bronx, New York
  - DelRicht Research, Charlotte, North Carolina
  - Eximia EquiHealth Research, LLC, Durham, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - West Clinical Research, Inc., Morehead City, North Carolina
  - OnSite Clinical Solutions, LLC, Salisbury, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Velocity Clinical Research - Cleveland, Beachwood, Ohio
  - Velocity Clinical Research - Springdale, Cincinnati, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Tekton Research, LLC, Edmond, Oklahoma
  - Lynn Health Science Institute East, Oklahoma City, Oklahoma
  - DelRicht Research, Tulsa, Oklahoma
  - Tekton Research, LLC, Yukon, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Central Erie Primary Care, Erie, Pennsylvania
  - Hatboro Medical Associates / Avacare, Horsham, Pennsylvania
  - DM Clinical Research, Philadelphia, Pennsylvania
  - DelRicht Research, Charleston, South Carolina
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Velocity Clinical Research - Spartanburg, Spartanburg, South Carolina
  - DelRicht Research, Hendersonville, Tennessee
  - DCT-HCWC, LLC dba Discovery Clinical Trials, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Lonestar Clinical Research, LLC, Dallas, Texas
  - Laguna Clinical Research Associates, LLC, Laredo, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Elevate Clinical Research, McAllen, Texas
  - Pearland Physicians, Pearland, Texas
  - Research Your Health, Plano, Texas
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas
  - Elevate Clinical Research, Seabrook, Texas
  - Javara, Inc., Stephenville, Texas
  - DM Clinical Research, Tomball, Texas
  - Cope Family Medicine / Avacare, Bountiful, Utah
  - Olympus Family Medicine / Avacare, Salt Lake City, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Rainier Clinical Research Center, Renton, Washington
- United Kingdom (30):
  - Queen Elizabeth Hospital, University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - Fylde Coast Clinical Research at Layton Medical Centre, Blackpool, England
  - Southmead Hospital, North Bristol NHS Trust - Clinical Research Centre, Bristol, England
  - Velocity Clinical Research - Bristol, Bristol, England
  - Eynsham Medical Centre, Eynsham, England
  - Velocity Clinical Research - High Wycombe, High Wycombe, England
  - HMC Health, The Meadows Centre for Health, The Great West Surgery, Hounslow, England
  - Leeds Teaching Hospitals NHS Trust - St. James's University Hospital, Leeds, England
  - University Hospitals of Leicester NHS Trust - Leicester Royal Infirmary, Leicester, England
  - hVIVO Services Limited, London, England
  - Panthera Enfield, London, England
  - Velocity Clinical Research - North London, London, England
  - North Manchester General Hospital, Manchester, England
  - The University of Nottingham Health Service, Nottingham, England
  - Wansford Research LTD, Peterborough, England
  - University Hospitals Plymouth NHS Trust, Plymouth, England
  - Panthera Preston, Preston, England
  - Panthera Rochdale, Rochdale, England
  - Velocity Clinical Research - Romford, Romford, England
  - Warrington and Halton Teaching Hospitals NHS Foundation Trust, Runcorn, England
  - Salford Royal Hospital, Salford, England
  - Panthera Sheffield, Sheffield, England
  - University Hospital Southampton NHS Foundation Trust, NIHR Southampton Clinical Research Facility, Southampton, England
  - Royal Cornwall Hospitals NHS Trust, Truro, England
  - Windrush Medical Practice, Witney, England
  - Panthera York, York, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - NHS Lothian - Western General Hospital, Edinburgh, Scotland
  - Queen Elizabeth University Hospital, Glasgow Clinical Research Facility, Glasgow, Scotland
  - Cardiff and Vale UHB - University Hospital of Wales, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: No